CLINICAL TRIAL: NCT01341145
Title: Physical Fitness, Cardiovascular and Brain Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Collaborators: American Federation for Aging Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010-04-0106; 8A0024 (Other Grant/Funding Number: American Federation for Aging Reseaerch)
Record Dates: First submitted 2011-03-30; First posted 2011-04-25 (Estimated); Last update posted 2014-04-14 (Estimated); Status verified 2014-04

CONDITIONS: Hypertension
Keywords: hypertension; aerobic exercise; relaxation; functional magnetic resonance imaging (fMRI); magnetic resonance spectroscopy (MRS); brain health
MeSH Terms: conditions — Hypertension | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aerobic Exersice (Experimental): 12-week moderate aerobic exercise program
  Interventions: Behavioral: Aerobic Exercise
- Relaxation (Active Comparator): 12-week at home progressive muscle relaxation program
  Interventions: Behavioral: Relaxation

INTERVENTIONS:
Behavioral: Aerobic Exercise — 12-week moderate-intensity aerobic exercise program designed in accordance with the recommended guidelines established by the American College of Sports Medicine
  Other Names: Exercise
  Arms: Aerobic Exersice
Behavioral: Relaxation — 12-week progressive muscle relaxation program (active control)
  Arms: Relaxation

SUMMARY:
The goal of this study is to determine if aerobic exercise or progressive muscle relaxation is associated with changes in cardiovascular health, brain function, and cognition.

DETAILED DESCRIPTION:
Cognition is the most important determinant of health status, quality of life and functional ability in older age. Therefore, early interventions that preserve and enhance cognitive function are crucial for ensuring successful aging. The most common treatable risk factor for late-life cognitive impairment is midlife hypertension (HTN). One highly promising intervention strategy is aerobic exercise as it has been associated cognitive benefits in non-demented older adults. However, it is still unclear whether this benefit is due simply to prevention of other risk factors (e.g., reductions in blood pressure) or if exercise can reverse the negative effects of HTN on the brain. The goals of the current study are to employ sensitive measures of neuroimaging and cognition in order to 1).Compare cerebral health in endurance trained versus sedentary middle aged adults with normal or borderline to stage 1 hypertension, 2). measure the effects of exercise training in previously sedentary middle aged adults adults with normal or borderline to stage 1 hypertension, and 3). examine if exercise-related differences and changes in neural integrity and cognition are mediated by systemic vascular health.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary adults Participants will be classified as sedentary if they have not engaged in regular physical exercise for at least one year prior to study enrollment.
* Ages 45-65
* Normal blood pressure or Borderline or stage 1 hypertension Borderline hypertension will be defined as systolic blood pressure between 120-139 mmHg and/or diastolic blood pressure between 80-89 mmHg. Stage 1 hypertension will be defined as systolic blood pressure between 140-159 mmHg and/or diastolic blood pressure between 90-99 mmHg.

Exclusion Criteria:

* Signs or symptoms of chronic heart disease
* Smoking (current or within the past 6 months)
* Peripheral artery disease (ankle-brachial index<0.9)
* Diabetes (fasting blood glucose>126 mg/L)
* Orthopedic problems that would prohibit participants from participating in exercise.
* Axis I psychiatric disorder
* Magnetic resonance contraindications
* Baseline Intellectual Quotient < 70
* Below chance performance on the practice items of the cognitive tasks
* Evidence of large vessel stroke on magnetic resonance imaging

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2011-03; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Percent signal change in Blood oxygen level-dependent (BOLD) response to a working memory task | change from baseline in blood oxygen level-dependent (BOLD) response to WM task at 14 weeks
  Blood oxygen level-dependent (BOLD) functional magnetic resonance imaging (fMRI) during 2-Back working memory task
N-acetyl aspartate (NAA) concentration | change from baseline in N-acetyl aspartate (NAA) concentration at 14 weeks
  Magnetic resonance spectroscopy (MRS) measurements of N-acetyl-aspartate (NAA)

CONTACTS AND LOCATIONS:
Overall Officials: Andreana Haley, PhD, Principal Investigator — University of Texas at Austin; Hirofumi Tanaka, Ph.D., Principal Investigator — University of Texas at Austin
Locations (1):
- University of Texas at Austin, Austin, Texas, United States